CLINICAL TRIAL: NCT00850512
Title: Study to Evaluate the Efficacy and Safety of Subsequent Treatment With the Zevalin (Ibritumomab Tiuxetan) in Elderly (More Than 60 Years) Patients With Diffuse Large B Cell Lymphoma After 4 Cycles of CHOP21-Rituximab (CHOP21-R) Therapy
Acronym: CHOP21+R-Z
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bologna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHOP21+R-Z
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibritumomab tiuxetan

ARMS (1):
- CHOP21 (Experimental): 4 cycles CHOP21-R plus Zevalin
  Interventions: Drug: CHOP21-R; Drug: Zevalin

INTERVENTIONS:
Drug: CHOP21-R — Four months for CHOP21-R and two treatment days one week apart
Drug: Zevalin — 12-week safety period for Zevalin

SUMMARY:
Study phase: Phase II Investigational product, dosage, and route of administration: Ibritumomab tiuxetan ("Zevalin) is composed of a murine IgG1 monoclonal antibody (ibritumomab) covalently bound to the chelating agent tiuxetan. To prepare the active therapeutic agent [90Y]-ibritumomab tiuxetan, the antibody is chelated with the β-emitter yttrium-90 chloride immediately before intravenous administration. Treatment with [90Y]-ibritumomab tiuxetan is preceded by an infusion of rituximab (Rituxan, Mabthera) in order to optimize the biodistribution of radiolabeled antibody by depleting CD20 positive B-cells. Rituximab is a chimeric human/murine IgG1 monoclonal antibody. The Zevalin study regimen is given as an infusion of rituximab 250 mg/m2 and (where biodistribution imaging or dosimetry is compulsory) 185 MBq (5mCi) of [111In]-ibritumomab tiuxetan on Day 1 followed 7 to 9 days later by a single dose of 14.8 MBq/kg (0.4 mCi/kg) of [90Y]-ibritumomab tiuxetan, maximal dose of 1184 MBq (32 mCi), preceded by 250 mg/m2 of rituximab.

Reference product, dosage, and route of administration: Not applicable Indication: stage II-IV diffuse large B-cell lymphoma (DLBCL) patients after 4 cycles of CHOP21-Rituximab (CHOP21-R) Study objectives: Evaluation of efficacy and safety of [90Y]-ibritumomab tiuxetan, as well as assessment of quality of life Patient population: Patients more than 60 years-of-age with DLBCL after 4 cycles of treatment with CHOP21-R Study design: Prospective, multicenter, open-label study designed to treat patients with a sequential front-line treatment represented by: 4 cycles CHOP21-R plus Zevalin Duration of treatment: Four months for CHOP21-R and two treatment days one week apart followed by a 12-week safety period for Zevalin Duration of study: Estimated duration of study is 18 months Methodology: Primary efficacy parameter: Overall response rate and complete response rate. Secondary efficacy parameters: Overall survival, disease-free survival, health-related quality of life. Safety parameters: Vital signs, adverse events (AEs), hematology, blood chemistry, and immunoglobulin levels Number of study centers: Planned total of 10 study centers in Italy Total number of patients, statistical rationale provided: Expected total of approximately 55 patients. The final sample size is based on the number of events observed for the primary efficacy endpoint as calculated in the sequential statistical model. Adverse events: AEs observed, mentioned upon open questioning and/or spontaneously reported will be documented.

Planned start and end of recruitment: Start of recruitment: 19/12/2006. End of recruitment: 04/11/2008.

Manufacturer(s) of the investigational /reference product(s): Ibritumomab tiuxetan is manufactured by Biogen IDEC, San Diego, CA and Cambridge, MA, USA. The isotopes yttrium-90 will be provided by European suppliers. There is no reference product in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, Ann Arbor stage II, III, or IV DLBCL according to the REAL/WHO classification (from initial diagnosis made prior to starting CHOP21-R therapy);
2. Central pathology review confirming the DLBCL diagnosis and CD20 positivity, and no evidence/evidence with an infiltration <25% of DLBCL in bone marrow;
3. The first part of the treatment of DLBCL must have been 4 cycles of standard CHOP21 chemotherapy (cyclophosphamide 750 mg/m2, doxorubicin 50 mg/m2, vincristine 1.4 mg/m2 up to a maximum of 2 mg on day 1, and at least 40 mg/m2/day prednisone on Days 1 to 5 every three weeks) in combination with rituximab (375 mg/m2);
4. Complete remission (CR), unconfirmed complete remission (CRu), partial response, and non-responder according to the International Workshop Response Criteria for NHL described by Cheson et al (18) after four cycles of CHOP21-R. CT scans of the neck, thorax, abdomen, and pelvis and PET total body must have been performed within 3 weeks after the last dose of the last course of CHOP21-R;
5. Patients 60-years-of-age or older at time of accrual;
6. WHO performance status (PS) of 0 to 2 within 1 week of accrual;
7. Absolute neutrophil count (ANC) more than 1.5 x 109/L within 1 week of accrual;
8. Hemoglobin (Hgb) more than 10 g/dL within 1 week of accrual;
9. Platelets more or equal than 150 x 109/L within 1 week of accrual.
10. Life expectancy of 3 months or longer
11. Written informed consent obtained according to local guidelines

Exclusion Criteria:

1. Presence of any other malignancy or history of prior malignancy except non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma;
2. Prior radioimmunotherapy, radiation therapy, or any other NHL therapy;
3. Presence of gastric, central nervous system (CNS), or testicular lymphoma at first diagnosis;
4. Histological transformation of low-grade NHL;
5. Known seropositivity for hepatitis C virus (HCV) or hepatitis B surface antigen (HbsAg);
6. Known history of HIV infection;
7. Abnormal liver function: total bilirubin > 1.5 x ULN or ALT > 2.5 x ULN within 1 week of accrual;
8. Abnormal renal function: serum creatinine > 2.0 x ULN within 1 week of accrual;
9. Nonrecovery from the toxic effects of CHOP21-R therapy;
10. Known hypersensitivity to murine or chimeric antibodies or proteins;
11. G-CSF or GM-CSF therapy within two weeks (or four weeks if pegylated) prior to screening laboratory sampling;
12. Concurrent severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months of study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study;
13. Treatment with investigational drugs less than 4 weeks before the planned Day 1 or nonrecovery from the toxic effects of such therapy;
14. Surgery less than 4 weeks before the planned Day 1 or nonrecovery from the side effects of such surgery;
15. Concurrent corticosteroid use for any reason except as premedication in case of known or suspected allergies to contrast media or as premedication for potential side effects of rituximab treatment;
16. Unwillingness or inability to comply with the protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)

PRIMARY OUTCOMES:
Overall response rate and complete response rate will be the primary endpoints

SECONDARY OUTCOMES:
overall survival (OS) and disease-free survival (DFS) will be the secondary endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto di Ematologia e Oncologia Medica Seràgnoli, Bologna, BO, Italy

REFERENCES:
- [Background] Zinzani PL, Tani M, Fanti S, Stefoni V, Musuraca G, Castellucci P, Marchi E, Farsad M, Fina M, Pellegrini C, Alinari L, Derenzini E, de Vivo A, Bacci F, Pileri S, Baccarani M. A phase II trial of CHOP chemotherapy followed by yttrium 90 ibritumomab tiuxetan (Zevalin) for previously untreated elderly diffuse large B-cell lymphoma patients. Ann Oncol. 2008 Apr;19(4):769-73. doi: 10.1093/annonc/mdm560. Epub 2008 Feb 25. PMID 18303033